CLINICAL TRIAL: NCT04087343
Title: Strength on Wheels: A Meal Delivery and Exercise Intervention for Homebound Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jessica Lee, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-19-0191; KL2TR003168 (NIH)
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Frailty
Keywords: homebound patients; exercise; nutrition
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Meals; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meals plus exercise (Experimental)
  Interventions: Behavioral: Meals plus exercise
- Meals only (Active Comparator)
  Interventions: Behavioral: Meals only

INTERVENTIONS:
Behavioral: Meals plus exercise — Patients will receive 12 weeks of meals on wheels meal delivery consisting of 3 meals per day during the weekdays with 6 frozen meals to cover the weekends.They will also receive an exercise kit on the first visit by the meal delivery driver with 2 tennis balls,2 1-pound hand weights, and one towel.Every week,the driver will give them 3 exercises from the National Institute on Aging's Go4Life Workout-to-Go book,1 exercise from each of 3 categories:strength/endurance, balance, and flexibility. They will be asked to do the 3 exercises every day.The meal delivery drivers will ask daily questions about physical activity and any potential injuries and the participants will be asked to track their own weekly exercise and physical activity as well as their monthly progress on a standardized log. All participants will also be asked to wear a fitness activity tracker which will monitor heart rate, activity level, and sleep habits for the duration of the study.
  Arms: Meals plus exercise
Behavioral: Meals only — Patients will receive 12 weeks of an enhanced meals on wheels (MOW) in-person meal delivery consisting of 3 meals per day (1 shelf-stable, 1 hot, and 1 frozen) during the weekdays (Monday through Friday) with 6 frozen meals at the end of the week to cover the weekends.The meal delivery drivers will ask daily questions about physical activity and any potential injuries and the participants will be asked to track their own weekly exercise and physical activity as well as their monthly progress on a standardized log. All participants will also be asked to wear a fitness activity tracker which will monitor heart rate, activity level, and sleep habits for the duration of the study.
  Arms: Meals only

SUMMARY:
The purpose of this study is to implement a home-based exercise program, administered through Interfaith Ministries of Greater Houston Meals on Wheels (MOWGH), and evaluate its effects on frailty status and nutritional markers in homebound older adults.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in UT-Health Harris Health House Call Program (HCP)
* Frail or pre frail by FFP
* medically stable

Exclusion Criteria:

* robust by FFP
* Mini-Cog score <3 and/or are unable to follow instructions
* pre-diagnosed terminal illness
* unable to ambulate,and/or are unable to use their upper extremities

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lee, MD,MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meals Only | Meals Plus Exercise
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meals Only | Meals Plus Exercise | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Frailty Status as Assessed by the Fried Frailty Phenotype (FFP) Screening Test.
Description: The FFP defines frailty as having 3 or more characteristics of unintentional weight loss, fatigue, decreased physical activity, weakness, and slowness.Those who have 1 or 2 characteristics are considered pre frail, while those who have no characteristics are robust.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Meals Only | Meals Plus Exercise
Number analyzed (Participants) | 4 | 5
Participants
  Frail | 2 | 2
  Prefrail | 2 | 3
  Robust | 0 | 0

2. Primary Outcome: Overall Frailty Status as Assessed by the Fried Frailty Phenotype (FFP) Screening Test.
Description: as for outcome 1
Time Frame: 12 weeks after study initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Meals Only | Meals Plus Exercise
Number analyzed (Participants) | 4 | 5
Participants
  Frail | 2 | 1
  Prefrail | 2 | 4
  Robust | 0 | 0

3. Secondary Outcome: Levels of Plasma Vitamin C
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ng/L | 2616.67 (2334.11) | 1180.56 (73.49)

4. Secondary Outcome: Levels of Plasma Vitamin C
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ng/L | 3738.89 (2714.39) | 2055.56 (304.29)

5. Secondary Outcome: Levels of Serum Folate
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ug/L | 20.32 (18.67) | 10.50 (1.52)

6. Secondary Outcome: Levels of Serum Folate
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ug/L | 19.56 (13.96) | 10.85 (3.57)

7. Secondary Outcome: Levels of Vitamin B12
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ng/L | 839.17 (593.41) | 575.83 (139.65)

8. Secondary Outcome: Levels of Vitamin B12
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ng/L | 875.42 (557.59) | 528.44 (160.04)

9. Secondary Outcome: Levels of Vitamin 25-OHD
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ug/L | 120.75 (93.16) | 86.41 (33.02)

10. Secondary Outcome: Levels of Vitamin 25-OHD
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
ug/L | 126.72 (120.6) | 61.68 (17.92)

11. Secondary Outcome: Levels of Methylmalonic Acid (MMA)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
pg/mL | 533.64 (420.41) | 406.93 (179.8)

12. Secondary Outcome: Levels of Methylmalonic Acid (MMA)
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
pg/mL | 554.55 (511.10) | 388.75 (161.44)

13. Secondary Outcome: Levels of Homocysteine (HCy)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pmol/uL
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
pmol/uL | 19.20 (3.93) | 18.21 (7.94)

14. Secondary Outcome: Levels of Homocysteine (HCy)
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Deviation); unit: pml/uL
Arm/Group | Meals Plus Exercise | Meals Only
Number analyzed (Participants) | 5 | 4
pml/uL | 18.83 (6.83) | 21.24 (5.81)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Meals Only | Meals Plus Exercise
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/5
Other Adverse Events (participants affected / at risk) | 2/4 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meals Only (N=4) | Meals Plus Exercise (N=5)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meals Only (N=4) | Meals Plus Exercise (N=5)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Poor Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Tooth Pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT04087343/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT04087343/ICF_001.pdf